CLINICAL TRIAL: NCT04611646
Title: Effects of Heat-suit Training on Training-associated Changes in Hemoglobin Mass, Muscle Characteristics and Endurance Performance in Elite Cyclists
Brief Title: Effects of Heat-suit Training on Biological and Performance Characteristics in Elite Cyclists
Acronym: HeatME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trainome 2020#025
Record Dates: First submitted 2020-10-20; First posted 2020-11-02 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-11

CONDITIONS: Heat-suit Endurance Training; Non-heat-suit Endurance Training
Keywords: Cycling; Heat; Hemoglobin mass; Skeletal muscle; Elite cyclists; Endurance performance; Mitochondria
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a five-week intervention. In the heat-suit arm, participants will conduct a 50-minute low-intensity cycling session with heat suit five time a week. In the none-heat-suit arm, participants will conduct similar amounts of low-intensity cycling without heat suit. These training sessions will complement the habitual training of the participants. Participants will be allocated into the two arms in a planned randomized manner. In short, participants will be stratified based on baseline performance levels (VO2max), whereby they will be allocated into the two intervention arms in a manner that ensures similar average performance levels between the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat-suit training (Experimental): Low-intensity endurance training with heat suit
  Interventions: Behavioral: Heat-suit endurance training
- Non-heat-suit training (Other): Low-intensity endurance training without heat suit
  Interventions: Behavioral: Non-heat-suit endurance training

INTERVENTIONS:
Behavioral: Heat-suit endurance training — Participants (elite cyclists) will conduct five 50-minute low-intensity cycling sessions with heat suit per week for five weeks. These sessions will complement their habitual training routines, which will consist of endurance training with intensities at or below lactate threshold. Participants will ingest 100 mg Fe2+ on a daily basis to support de novo synthesis of hemoglobin
  Other Names: Heat training
  Arms: Heat-suit training
Behavioral: Non-heat-suit endurance training — Participants (elite cyclists) will conduct low-intensity cycling without heat suit for five weeks (volume- and intensity-matched to the heat-suit arm). Participants will ingest 100 mg Fe2+ on a daily basis to support de novo synthesis of hemoglobin
  Other Names: Control group
  Arms: Non-heat-suit training

SUMMARY:
The overall objective of the study is to investigate the effects of five weeks of heat-suit training on training-associated changes in hemoglobin mass, skeletal muscle characteristics and endurance exercise performance in elite cyclists

DETAILED DESCRIPTION:
Endurance exercise performance depends on a range of determinants, including hemoglobin mass in blood and content of respiratory mitochondria in skeletal muscle. Low-intensity training (LIT) with heat exposure may be beneficial for development of these variables. The purpose of this study is to investigate the effects of five weeks of LIT-training with heat suit (five times a week; 50 min per session) on hemoglobin mass and other blood characteristics in elite cyclists (males and females) compared to a non-heat-suit training control group, including subsequent investigation of the retrograde effects of ~one month of training without heat suit. The study will also investigate the effects of heat-suit training on endurance exercise performance/performance determinants and other muscle biological charateristics, and will investigate the basic characteristics of mitochondrial function and abundances in these highly trained athletes. Training sessions with heat suit (or lack thereof) will complement the habitual training routines of the participants.

ELIGIBILITY:
Inclusion Criteria:

* VO2max > 65 ml/kg/min (male participants)
* VO2max > 50 ml/kg/min (female participants)
* >7 hours of endurance training per week for the 6 months leading up to the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Hemoglobin mass | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Hemoglobin mass measured using CO rebreathing (g)

SECONDARY OUTCOMES:
Maximal oxygen consumption | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Maximal oxygen consumption measured during an incremental cycling exercise test to exhaustion
Maximal aerobic power output | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Maximal aerobic power output measured as mean power output during the last minute of an incremental cycling exercise test to exhaustion
Power output at lactate threshold | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Power output at 4 mmol blood lactate concentration measured during an incremental cycling exercise test (with 5 minute steps)
Gross efficiency | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Contribution of total energy turnover to power output in the fresh and fatigued state
Fractional utilization of VO2max (incremental test) | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Fractional utilization of VO2max measured at 4 mmol blood lactate concentrations measured during an incremental cycling exercise test (with 5 minute steps)
Fractional utilization of VO2max (15-minute performance test) | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Fractional utilization of VO2max measured during a 15-minute performance test
Sprint performance | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Mean power output measured during a 10-second all-out cycling sprint
Performance during a 15-minute all-out cycling test | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Mean power output measured during a 15-minute all-out cycling test
Performance during a 40-minute all-out cycling test | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Mean power output measured during a 40-minute all-out cycling test
Maximal concentric force production | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Maximal concentric force production measured using a seated leg press test
Gene expression in skeletal muscle | Changes from before the intervention (T0) to immediately after the intervention (T1)
  RNA abundances in m. vastus lateralis measured using qPCR (e.g. messenger RNA and ribosomal RNA)
Mitochondrial respiration in skeletal muscle | Immediately after the intervention (T1)
  The ability of muscle mitochondria (extracted from homogenate; m. vastus lateralis) to consume oxygen in vitro
Mitochondrial content in skeletal muscle | Immediately after the intervention (T1)
  Mitochondria content in m. vastus lateralis measured using electron microscopy
Total RNA content in skeletal muscle | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Total RNA content in m. vastus lateralis (per unit tissue weight) measured using spectrophotometry
Blood volume | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Blood volume measured using CO rebreathing
Plasma volume | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Plasma volume measured using CO rebreathing
Red blood cell volume | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Red blood cell volume measured using CO rebreathing
Hematocrit | Changes from before the intervention (T0) to immediately after the intervention (T1)
  Hematocrit measured using centrifugation
Hemoglobin mass | Changes from immediately after the intervention (T1) to one month after the intervention (T2)
  Hemoglobin mass measured using CO rebreathing (g)
Blood volume | Changes from immediately after the intervention (T1) to one month after the intervention (T2)
  Blood volume measured using CO rebreathing
Plasma volume | Changes from immediately after the intervention (T1) to one month after the intervention (T2)
  Plasma volume measured using CO rebreathing
Red blood cell volume | Changes from immediately after the intervention (T1) to one month after the intervention (T2)
  Red blood cell volume measured using CO rebreathing
Hematocrit | Changes from immediately after the intervention (T1) to one month after the intervention (T2)
  Hematocrit measured using centrifugation

OTHER OUTCOMES:
Training volume | Throughout study completion (daily), an average of five weeks
  Self-reported training volume measured as time-spent in different exercise intensity zones
Iron intake | Throughout study completion (daily), an average of five weeks
  Self-reported intake of iron supplements

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Lofthus, Study Chair — Research Administrator
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Inland Norway, Norway